CLINICAL TRIAL: NCT02084641
Title: Adipose Tissue Response to Overfeeding in Insulin Resistance-Prone vs. Insulin Sensitive Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Tracey McLaughlin, Associate Professor, Stanford University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20281
Record Dates: First submitted 2013-03-12; First posted 2014-03-12 (Estimated); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Insulin Resistance; Obesity
Keywords: ectopic fat; obesity; triglyceride storage; adipocyte; overfeeding; intrahepatic fat; adipocyte proliferation; inflammation; macrophage
MeSH Terms: conditions — Insulin Resistance; Obesity; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Insulin resistant (Experimental): Both groups will be given the same intervention and then outcomes compared between groups
  Interventions: Other: Over feeding
- Insulin Sensitive (Experimental): Both groups will be given the same intervention and then outcomes compared between groups
  Interventions: Other: Over feeding

INTERVENTIONS:
Other: Over feeding — Study participants will be given low saturated fat snacks, an additional 750-1000 calories to gain 6-8 lbs over 4 weeks

SUMMARY:
Obesity has become an epidemic worldwide. Data from our laboratory and others demonstrate that most of the excess morbidity from obesity is related to insulin resistance (IR). While total adiposity correlates with insulin resistance, not all obese individuals are IR. When obese IR individuals lose weight in response to caloric restriction, even moderate loss of body fat results in improved insulin sensitivity (IS). With massive weight loss, either dietary or surgical, even the most IR individuals can completely reverse their insulin resistance. But why is one individual IR at a BMI of 26 and another IS at a BMI of 35? There must be differences in the manner in which adipose cells/tissue respond to caloric excess and weight gain. One potentially unifying hypothesis with regard to obesity-associated insulin resistance is that those individuals who fail to respond to caloric excess/obesity with adequate adipocyte differentiation and expanded subcutaneous fat storage capacity develop increased circulating FFAs, ectopic fat deposition, stress on adipocytes, triggering localized and systemic inflammation and ultimately insulin resistance in skeletal muscle.

Clearly, the best way to examine the human response to obesity is to challenge overweight individuals with the need to store excess triglyceride in adipose tissue. Specific aims are:

1. Test the hypothesis that impaired adipogenesis and fat storage capacity are associated with insulin resistance by comparing 1) cell size distribution; 2) gene markers of adipose cell differentiation; 3) differentiation of isolated preadipocytes in IR-prone vs IS individuals subjected to caloric excess.
2. Determine if circulating (daylong FFA, two-stage Insulin Suppression Test) and ectopic fat (MRI liver, CT abdomen) are worsened to a greater degree in IR-prone vs IS individuals subjected to caloric excess.
3. Determine whether differences in inflammation and/or innate or adaptive immune response are associated with insulin resistance by comparing differences in resident dendritic cells, macrophages and their activation profiles, changes in T-cell subpopulations, and other inflammatory mediators in IR-prone vs IS individuals who are subjected to caloric excess via overfeeding.
4. Exploratory: Evaluate IR-prone vs IS individuals for evidence of hypoxia and insufficient angiogenic response in response to caloric excess.

ELIGIBILITY:
Inclusion Criteria:

* BMI 25-35 kg/m2
* Healthy adults
* Age 35-65
* Weight stable
* Nondiabetic

Exclusion Criteria:

* Major organ disease such as heart, kidney, liver
* Malignancy
* Inflammatory conditions (eg. lupus, rheumatoid arthritis, Crohn's disease)
* Eating disorder h/o bariatric surgery or liposuction use of blood thinners such as Coumadin (aspirin is ok)

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2011-09 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Subcutaneous adipose cell triglyceride storage capacity/differentiation | 3 years
  this will be quantified by measuring: 1) adipose cell size distribution; 2) gene markers of adipose cell differentiation; 3) differentiation of isolated preadipocytes in IR-prone vs IS individuals subjected to caloric excess; in vivo triglyceride synthesis using stable isotope methods

SECONDARY OUTCOMES:
Ectopic fat | 3 years
  Fat deposited in liver (MRI), visceral (intraabdominal) abdominal (CT) versus subcutaneous abdominal and thigh fat (CT)

OTHER OUTCOMES:
Adipose tissue and systemic inflammation: both innate or adaptive immune response | 3 years
  Flow cytometry will be used to quantitate, in both adipose tissue and plasma, populations of dendritic cells, T-cell subpopulations, and macrophages

CONTACTS AND LOCATIONS:
Overall Officials: Tracey McLaughlin, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States